CLINICAL TRIAL: NCT02025712
Title: A Phase II Open-label Pilot Study Evaluating the Maintenance Therapy With Exemestane Plus Everolimus After Induction Chemotherapy in Patients With Hormone-receptor Positive Metastatic Breast Cancer
Brief Title: Exemestane Plus Everolimus for Hormone-receptor Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Organisation for Oncology and Translational Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M004/EXE-EVE
Record Dates: First submitted 2013-12-16; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast
MeSH Terms: interventions — exemestane; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exemestane plus Everolimus (Experimental): Exemestane 25 mg daily in combination with Everolimus 10 mg daily until disease progression or intolerable toxicity
  Interventions: Drug: Exemestane; Drug: Everolimus

INTERVENTIONS:
Drug: Exemestane — Commercially available exemestane was supplied to sites as 25-mg tablets according to local regulations.
  Other Names: Aromasin
Drug: Everolimus — Everolimus was administered by continuous oral dosing of two 5-mg tablets or one 10-mg tablets.
  Other Names: Afinitor, RAD001

SUMMARY:
The purpose of this study is to determine whether exemestane plus everolimus are effective in the treatment of patients who have achieved disease stabilization after induction chemotherapy for hormone-receptor positive metastatic breast cancer.

DETAILED DESCRIPTION:
Postmenopausal women with HR-positive, HER2-negative metastatic breast cancer achieving clinical benefit after the induction chemotherapy for visceral disease with sign(s) and/or symptom(s) will be recruited to receive study the maintenance treatment of everolimus plus exemestane.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women as defined in the protocol page 9;
* Histologically and/or cytologically confirmed invasive breast cancer with stage IV disease according to AJCC;
* Confirmed ER/PR-positive, and HER-2 negative tumor;
* Disease progression on or following prior endocrine therapy with tamoxifen or non-steroidal aromatase inhibitor, as defined in protocol, prior to standard of care (SOC) induction chemotherapy
* Patient with documented evidence of visceral disease (including but not limited to hepatic involvement and pulmonary lymphangitic spread of tumor) with sign(s) and/or symptom(s) prior to SOC induction chemotherapy should achieve disease stabilization after the SOC induction chemotherapy, confirmed upon 2 consecutive routine tumor assessments;
* ECOG performance status ≤ 2 or Karnofsky performance status ≥ 50% prior to the start of study treatment;
* Adequate organ function prior to the start of study treatment as defined in the protocol;
* Able to swallow and retain oral medication;
* Able to give written informed consent;

Exclusion Criteria:

* Male patient;
* Metastatic disease limited to the bone or soft tissues only and with no history of other visceral metastases;
* History of brain or other CNS metastases;
* Previous treatment with exemestane, unless exemestane was administered in the adjuvant setting and stopped >1 year before metastatic relapse;
* Untreated with SOC chemotherapy for invasive breast cancer with stage IV disease according to AJCC - or - treated with SOC chemotherapy for invasive breast cancer with stage IV disease according to AJCC without clinical benefit;
* History of neurological or psychiatric disorders;
* Any serious cardiovascular diseases in the previous 6 months;
* Impairment of gastrointestinal function or gastrointestinal disease;
* Patients with uncontrolled infection;
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin defined as 1 mg a day);
* Chronic treatment with systemic steroids or another immunosuppressive agent;
* Patients with a pre-existing peripheral neuropathy > grade 1;
* Patients who are hepatitis B and/or hepatitis C carriers;
* Known human immunodeficiency virus infection;
* Prior exposure to mTOR inhibitors;
* Hypersensitivity to rapamycin or other similar compounds;
* Patients taking medications known to be inhibitors or inducers of CYP3A4 and/or PgP will not be included in this study;
* Prior treatment with any investigational agent within the preceding 4 weeks;
* Other conditions in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Every 8 weeks in the first 24 weeks of treatment and every 12 weeks thereafter, up to 8 months (estimated)
  defined as from date of treatment initiation with everolimus plus exemestane to the date of progression or death if no documented disease progression

SECONDARY OUTCOMES:
Response rate | Every 8 weeks, up to 8 months (estimated)
Clinical benefit rate | Every 8 weeks, up to 8 months (estimated)
Overall survival | date of treatment initiation with everolimus plus exemestane until the date of death, censored at the last date known alive, whichever came first, assessed up to 32 months
Incidence of Adverse Events (AEs)/Serious Adverse Events (SAEs) | Continuous during the study, up to 28 days after the last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Louis Chow, Principal Investigator — Organisation for Oncology and Translational Research
Locations (1):
- Unimed Medical Institute, Hong Kong, China